CLINICAL TRIAL: NCT06507800
Title: Cancer as a complicATion in reCipients of Autologous Hematopoietic Stem Cell Transplantation for Autoimmune Disease iNdiCation trEated in FRance and Canada?
Acronym: CATCH CANCER
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231300
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Autoimmune Diseases
Keywords: Autoimmune diseases; Hematopoietic Stem Cell Transplantation; Cancer
MeSH Terms: conditions — Autoimmune Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MATHEC cohort: French national registry of patients treated by Autologous haematopoietic stem cell transplantation (AHSCT) for their autoimmune disease
  Interventions: Other: Observational cohort
- Ottawa cohort: Patients treated by AHSCT for their autoimmune disease and followed in Ottawa Hospital
  Interventions: Other: Observational cohort
- Calgary cohort: Patients treated by AHSCT for their autoimmune disease and followed in Calgary Hospital
  Interventions: Other: Observational cohort

INTERVENTIONS:
Other: Observational cohort — Cancer incidence after AHSCT for an autoimmune indication.

SUMMARY:
Autologous Hematopoietic Stem Cell Transplantation (AHSCT) is a treatment option for several types of Autoimmune Disease (AD) in patients who remain active despite disease modifying therapies. In this setting, AHSCT was shown to improve overall survival, event free survival and quality of life, with a grade A level evidence for systemic sclerosis (SSc) and multiple sclerosis (MS) patients and its benefit varies according to the AD type and the patient status for the other indications. The number of AHSCT for AD has increased in the past twenty years at each country level in Europe and also in Canada.

Information about cancer after AHSCT for AD is scant, although the AD patients population per se has an increased rate of cancer. This cancer risk can be explained in part by the long term use of immunosuppressive drugs or by other risk factors related to the AD (as in SSc or Crohn) or to the patient. In addition to pretransplant potential risk factors for cancer in AD patients, the use of conditioning regimen, which may vary from low, medium or high immunosuppressive to myeloablative chemotherapy when irradiation is added to the proecedure, may favor the onset of cancer after AHCST. Updated analysis and review of the literature until march 2023 led us to identify only twenty-two cases of cancer or hematological malignancies reported after AHSCT recipients for an AD.

The incidence of cancer after AHSCT for AD was never considered as a primary endpoint in any previous study.

In this context, the aim of this study is to describe the incidence of cancer after autologous hematopoietic stem cell transplantation (AHSCT) for auto-immune diseases (AD) in the French MATHEC (French scientific network for AD and cellular therapies) and the Ottawa and Calgary patients cohorts from Day 0 until twenty years follow up after AHSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years at AHSCT
2. Underwent first AHSCT for any AD indication
3. Included in the French MATHEC-SFGM-TC registry or the Canadian Ottawa and Calgary databases
4. AHSCT between January, 1st, 2000 and December, 31st, 2022
5. Informed consent for data registration in the respective original registry/database

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated bu AHSCT for their autoimmune disease, and followed either in France (MATHEC registry), Calgary (Canada) or Ottawa (Canada)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of any cancer after AHSCT for an autoimmune indication | Up to 22 years after AHSCT
  Description of the cancers by site according to the International Classification of Diseases for Oncology, 3rd Edition

SECONDARY OUTCOMES:
Cumulative incidence of cancer by age and sex | Up to 22 years after AHSCT
Incidence of Non-relapse mortality (NRM) | Up to 22 years after AHSCT
Incidence of disease relapse/progression | Up to 22 years after AHSCT
Overall survival (OS) | Up to 22 years after AHSCT
Causes of death (Causes of death will be classified as related to primary AD disease, the secondary cancer or any other cause). | Up to 22 years after AHSCT

IPD SHARING:
Plan to Share IPD: Undecided